CLINICAL TRIAL: NCT02914964
Title: Dietary Approaches to Treat Multiple Sclerosis-Related Fatigue Study
Acronym: Waves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 201604705
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Fatigue; Quality of Life; Diet
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swank Diet (Experimental): Individuals randomized to this arm will follow a low saturated fat diet starting at week 12.
  Interventions: Behavioral: Swank Diet
- Wahls Elimination Diet (Experimental): Individuals randomized to this arm will follow a modified paleolithic diet that eliminates all grains, dairy, eggs, legumes, and nightshade vegetables/spices starting at week 12.
  Interventions: Behavioral: Wahls Elimination Diet

INTERVENTIONS:
Behavioral: Swank Diet — A Registered Dietitian Nutritionist (RDN) skilled in motivational interviewing will provide nutrition counseling to study participants to assist them in following the Swank Diet at home. An in-person counseling session will occur at study visits 2 and 3. Five telephone counseling calls will occur between visits 2 and 3. The study participant may contact the RDN with questions at any time during the intervention.
  Arms: Swank Diet
Behavioral: Wahls Elimination Diet — A Registered Dietitian Nutritionist (RDN) skilled in motivational interviewing will provide nutrition counseling using to study participants to assist them in following the Wahls Elimination Diet at home. An in-person counseling session will occur at study visits 2 and 3. Five telephone counseling calls will occur between visits 2 and 3. The study participant may contact the RDN with questions at any time during the intervention.
  Arms: Wahls Elimination Diet

SUMMARY:
The purpose of this study is to compare the effect of the Swank Diet (low saturated fat) and the Wahls Elimination Diet (modified paleo) on fatigue levels in individuals with relapsing-remitting multiple sclerosis who have documented fatigue. Participants will follow their usual diet for 12 weeks and then be randomly assigned to follow one of the two diets for 24 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effect of the Swank Diet (low saturated fat) and the Wahls Elimination Diet (modified paleo) on fatigue levels in individuals with relapsing-remitting multiple sclerosis who have documented fatigue. Participants will follow their usual diet for 12 weeks and then be randomly assigned to follow one of the two diets for 24 weeks. Individuals will continue with their current treatments in addition to following the study diet.

The study requires four visits to the University of Iowa Hospitals and Clinics in Iowa City, Iowa. Visits will be 12 weeks apart. Study activities include fasting blood draws, weighed food records, motor and cognitive testing, physical activity assessment, questionnaires, and daily diet checklists while following the study diet. Some reimbursement available.

ELIGIBILITY:
Inclusion Criteria:

* Willing to allow your neurologist to sign a letter confirming multiple sclerosis diagnosis and criteria used in diagnosis
* Relapsing-Remitting Multiple Sclerosis as documented by the McDonald Criteria confirmed by their treating neurologist
* Fatigue as documented by a Fatigue Severity Scale score of greater than or equal to 4
* Between the ages of 18 and 70
* Body Mass Index greater than or equal to 19
* Ability to shop for and prepare or have someone in the family shop for and prepare home cooked meals according to study diet guidelines
* Willingness to keep detailed food records
* Willing to eat a diet that includes more vegetables and excludes many comfort foods such as those made with white flour,
* Willing to eat a diet that eliminates red meat (beef, pork, lamb, veal) and saturated fats (butter, coconut oil, margarine, hydrogenated oils found in processed foods) to 1 tablespoon per day
* Must not be pregnant or planning to become pregnant in the next year
* Willing to eat meat (eg, chicken, turkey, fish)
* Willingness to follow either the Wahls Elimination diet or the Swank diet
* Individuals who have had gastric bypass surgery have obtained a signed statement from their physician indicating they are weight stable and a suitable candidate for this study
* Normal or mild cognitive impairment as measured by the Short Portable Mental Status Questionnaire
* Willing to have blood drawn
* Be able to walk 25 feet without support, or with only unilateral support (i.e. cane in one hand)

Exclusion Criteria:

* Taking insulin or Coumadin
* Relapse within past 12 weeks
* Treatment for a cancer (other than skin cancer) currently or in the prior 12 months
* Diagnosis of heart failure, liver cirrhosis, angina, history of kidney stones, psychiatric disease likely to make adherence to the study interventions more difficult including eating disorders, but excluding depression and anxiety
* Body Mass Index less than 19
* Moderate to severe mental impairment as measured by the Short Portable Mental Status questionnaire
* Inability to shop for and prepare home cooked meals by the subject or a companion
* Unwillingness to eat meat
* Participation in another research study that involves multiple sclerosis or other medications, diet, supplement, exercise or other treatments
* Inability to keep food records with sufficient detail to asses dietary intake or complete study questionnaires
* Unwilling to have blood drawn
* Pregnant or planning to become pregnant in the next year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Change in participant perceived fatigue severity | 12-24 weeks
  Participant questionnaire asking about fatigue: Fatigue Severity Scale score - a 9-questions scale ranging from 1 (complete disagreement with the question) to 7 (complete agreement with the questions)
Change in participant perceived fatigue severity | 12-36 weeks
  Participant questionnaire asking about fatigue: Fatigue Severity Scale score - a 9-questions scale ranging from 1 (complete disagreement with the question) to 7 (complete agreement with the questions)
Change in the impact of fatigue on daily life | 12-24 weeks
  Modified Fatigue Impact Scale score: Participant questionnaire asking about impact of fatigue impact daily life: Modified Fatigue Impact Scale score. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The MFIS consists of 21 items. Scoring is based upon a sum of the responses. Total score ranges from 0 to 84.
Change in the impact of fatigue on daily life | 12-36 weeks
  Modified Fatigue Impact Scale score: Participant questionnaire asking about impact of fatigue impact daily life: Modified Fatigue Impact Scale score. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The MFIS consists of 21 items. Scoring is based upon a sum of the responses. Total score ranges from 0 to 84.

SECONDARY OUTCOMES:
Change in participant walk speed | 12-24 weeks
  6 Minute Walk Test
Change in participant walk speed | 12-36 weeks
  6 Minute Walk Test
Change in gait (walk) | 12-24 weeks
  25 foot Walk Test
Change in gait (walk) | 12-36 weeks
  25 foot Walk Test
Change in fine motor function | 12-24 weeks
  Pegboard test
Change in fine motor function | 12-36 weeks
  Pegboard test
Change in nutrient intake based on the recommended daily allowance (RDA) | 12-24 weeks
  Nutrient intake calculated from 3-day weighed food records and Food Frequency Questionnaire and Participant blood measurements of insulin, glucose, hemoglobin A1C, Vitamin K, homocysteine, lipids, fatty acid profile and vitamin D.
Change in nutrient intake based on the recommended daily allowance (RDA) | 12-36 weeks
  Nutrient intake calculated from 3-day weighed food records and Food Frequency Questionnaire and Participant blood measurements of insulin, glucose, hemoglobin A1C, Vitamin K, homocysteine, lipids, fatty acid profile and vitamin D.
Change in cognitive function | 12-24 weeks
  Symbol Digit Modalities Test - oral. An oral test of sequencing symbols. •Participant substitutes a number for meaningless geometric shapes based on a key that assigns a specific number to each shape. Scoring is based on the number of correct substitutions.
Change in cognitive function | 12-36 weeks
  Symbol Digit Modalities Test - oral. An oral test of sequencing symbols. •Participant substitutes a number for meaningless geometric shapes based on a key that assigns a specific number to each shape. Scoring is based on the number of correct substitutions.
Change in steps per day | 12-24 weeks
  Measured by accelerometer
Change in steps per day | 12-36 weeks
  Measured by accelerometer
Change in participant Quality of Life (QoL) - General Health | 12-24 weeks
  Multiple Sclerosis 54 Quality of Life Questionnaire. A series of questions about quality of life and social functioning. Score 0 to 100.
Change in participant Quality of Life (QoL) - General Health | 12-36 weeks
  Multiple Sclerosis Quality of Life Questionnaire. A series of questions about quality of life and social functioning. Score 0 to 100.
Change in participant Quality of Life (QoL) - Mental Health | 12-24 weeks
  Multiple Sclerosis Quality of Life Questionnaire A series of questions about quality of life and social functioning. Score 0 to 100.
Change in participant Quality of Life (QoL) - Mental Health | 12-36 weeks
  Multiple Sclerosis Quality of Life Questionnaire A series of questions about quality of life and social functioning. Score 0 to 100.
Change in total sleep time | 12-24 weeks
  Total sleep time is measured in hours and minutes and tracked by accelerometer worn by participants throughout the study
Change in total sleep time | 12-36 weeks
  Total sleep time is measured in hours and minutes and tracked by accelerometer worn by participants throughout the study
Change in perceived anxiety | 12-24 weeks
  Perceived anxiety is measured by the Hospital Anxiety and Depression Scale (HADS), a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence.
Change in perceived anxiety | 12-36 weeks
  Perceived anxiety is measured by the Hospital Anxiety and Depression Scale (HADS), a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence.
Change in perceived depression | 12-24 weeks
  Perceived depression is measured by the Hospital Anxiety and Depression Scale (HADS), a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence.
Change in perceived depression | 12-36 weeks
  Perceived depression is measured by the Hospital Anxiety and Depression Scale (HADS), a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, MBA, Principal Investigator — University of Iowa; Linda Snetselaar, PhD, RD,, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisht B, Darling WG, Shivapour ET, Lutgendorf SK, Snetselaar LG, Chenard CA, Wahls TL. Multimodal intervention improves fatigue and quality of life in subjects with progressive multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2015;5:19-35. doi: 10.2147/DNND.S76523. Epub 2015 Feb 27. PMID 30728736
- [Background] Bisht B, Darling WG, Grossmann RE, Shivapour ET, Lutgendorf SK, Snetselaar LG, Hall MJ, Zimmerman MB, Wahls TL. A multimodal intervention for patients with secondary progressive multiple sclerosis: feasibility and effect on fatigue. J Altern Complement Med. 2014 May;20(5):347-55. doi: 10.1089/acm.2013.0188. Epub 2014 Jan 29. PMID 24476345
- [Background] SWANK RL. Multiple sclerosis; a correlation of its incidence with dietary fat. Am J Med Sci. 1950 Oct;220(4):421-30. No abstract available. PMID 14771073
- [Background] SWANK RL. Treatment of multiple sclerosis with a low-fat diet. J Am Diet Assoc. 1960 Apr;36:322-5. No abstract available. PMID 13836031
- [Background] SWANK RL. Treatment of multiple sclerosis with low-fat diet. AMA Arch Neurol Psychiatry. 1953 Jan;69(1):91-103. doi: 10.1001/archneurpsyc.1953.02320250097011. No abstract available. PMID 12996138
- [Background] SWANK RL. Treatment of multiple sclerosis with low-fat diet; results of five and one-half years' experience. AMA Arch Neurol Psychiatry. 1955 Jun;73(6):631-44. doi: 10.1001/archneurpsyc.1955.02330120035004. No abstract available. PMID 14375427
- [Background] SWANK RL. Treatment of multiple sclerosis with low-fat diet: result of seven years' experience. Ann Intern Med. 1956 Nov;45(5):812-24. doi: 10.7326/0003-4819-45-5-812. No abstract available. PMID 13373189
- [Background] Swank RL. Multiple sclerosis: twenty years on low fat diet. Arch Neurol. 1970 Nov;23(5):460-74. doi: 10.1001/archneur.1970.00480290080009. No abstract available. PMID 5471652
- [Background] Swank RL. Multiple sclerosis: fat-oil relationship. Nutrition. 1991 Sep-Oct;7(5):368-76. PMID 1804476
- [Background] SWANK RL, BOURDILLON RB. Multiple sclerosis: assessment of treatment with a modified low-fat diet. J Nerv Ment Dis. 1960 Dec;131:468-88. No abstract available. PMID 13774215
- [Background] Swank RL, Dugan BB. Effect of low saturated fat diet in early and late cases of multiple sclerosis. Lancet. 1990 Jul 7;336(8706):37-9. doi: 10.1016/0140-6736(90)91533-g. PMID 1973220
- [Background] Swank RL, Goodwin J. Review of MS patient survival on a Swank low saturated fat diet. Nutrition. 2003 Feb;19(2):161-2. doi: 10.1016/s0899-9007(02)00851-1. No abstract available. PMID 12591551
- [Background] Swank RL, Goodwin JW. How saturated fats may be a causative factor in multiple sclerosis and other diseases. Nutrition. 2003 May;19(5):478. doi: 10.1016/s0899-9007(02)01099-7. No abstract available. PMID 12714108
- [Result] Shemirani F, Titcomb TJ, Saxby SM, Eyck PT, Rubenstein LM, Hoth KF, Snetselaar LG, Wahls TL. Association of serum homocysteine, folate, and vitamin B12 and mood following the Swank and Wahls elimination dietary interventions in relapsing-remitting multiple sclerosis: Secondary analysis of the WAVES trial. Mult Scler Relat Disord. 2023 Jul;75:104743. doi: 10.1016/j.msard.2023.104743. Epub 2023 May 1. PMID 37148578
- [Result] Crippes LJ, Saxby SM, Shemirani F, Bisht B, Gill C, Rubenstein LM, Ten Eyck P, Carr LJ, Darling WG, Hoth KF, Kamholz J, Snetselaar LG, Titcomb TJ, Wahls TL. Diet-induced changes in functional disability are mediated by fatigue in relapsing-remitting multiple sclerosis: A secondary analysis of the WAVES randomized parallel-arm trial. Mult Scler J Exp Transl Clin. 2023 Oct 30;9(4):20552173231209147. doi: 10.1177/20552173231209147. eCollection 2023 Oct-Dec. PMID 37916030
- [Result] Villa AT, Tu BH, Titcomb TJ, Saxby SM, Shemirani F, Ten Eyck P, Rubenstein LM, Snetselaar LG, Wahls TL. Association between improved metabolic risk factors and perceived fatigue during dietary intervention trial in relapsing-remitting multiple sclerosis: A secondary analysis of the WAVES trial. Front Neurol. 2023 Jan 19;13:1022728. doi: 10.3389/fneur.2022.1022728. eCollection 2022. PMID 36742040
- [Result] Wahls TL, Titcomb TJ, Bisht B, Eyck PT, Rubenstein LM, Carr LJ, Darling WG, Hoth KF, Kamholz J, Snetselaar LG. Impact of the Swank and Wahls elimination dietary interventions on fatigue and quality of life in relapsing-remitting multiple sclerosis: The WAVES randomized parallel-arm clinical trial. Mult Scler J Exp Transl Clin. 2021 Jul 31;7(3):20552173211035399. doi: 10.1177/20552173211035399. eCollection 2021 Jul-Sep. PMID 34377527
- [Derived] Wahls T, Scott MO, Alshare Z, Rubenstein L, Darling W, Carr L, Smith K, Chenard CA, LaRocca N, Snetselaar L. Dietary approaches to treat MS-related fatigue: comparing the modified Paleolithic (Wahls Elimination) and low saturated fat (Swank) diets on perceived fatigue in persons with relapsing-remitting multiple sclerosis: study protocol for a randomized controlled trial. Trials. 2018 Jun 4;19(1):309. doi: 10.1186/s13063-018-2680-x. PMID 29866196